CLINICAL TRIAL: NCT01587937
Title: Hospital Wide Roll-Out of Antimicrobial Stewardship: A Stepped Wedge Randomized Controlled Trial
Brief Title: Hospital Wide Roll-Out of Antimicrobial Stewardship
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 416-2009
Record Dates: First submitted 2012-04-13; First posted 2012-04-30 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Bacterial Infections
Keywords: Antibiotic stewardship.; Clostridium difficile infection.; Antibiotic resistance.
MeSH Terms: conditions — Bacterial Infections; Clostridium Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antibiotic stewardship intervention (Experimental): Audit-and-feedback intervention to prescribers of patients receiving 3rd or 10th day of targeted broadspectrum antimicrobial
  Interventions: Other: Antibiotic stewardship audit-and-feedback to prescribers of patients receiving 3rd or 10th day of targeted broadspectrum antibiotics
- Control (No Intervention): The pre-intervention period will serve as the control period on each medical and surgical service. The cross-over is uni-directional from control to intervention; all services receive the intervention by the end of the study. This is a stepped wedge design. The order of roll-out is randomized.

INTERVENTIONS:
Other: Antibiotic stewardship audit-and-feedback to prescribers of patients receiving 3rd or 10th day of targeted broadspectrum antibiotics — See primary outcome for list of targeted drugs. See citations for previous publications describing the intervention.
  Arms: Antibiotic stewardship intervention

SUMMARY:
Dramatic increases in antibiotic utilization in hospitals continue to drive antibiotic resistance among hospital-acquired pathogens. However, 30-50% of the antibiotic use in hospitals is unnecessary or inappropriate. The Infectious Diseases Society of America has published guidelines stating that all hospitals should develop an institutional program to enhance antimicrobial stewardship. At Sunnybrook Health Sciences Centre, an antibiotic stewardship audit-and-feedback intervention for all patients reaching their third or tenth day of broadspectrum antibiotic use in intensive care, resulted in a reduction of antibiotic use, antibiotic costs, and Clostridium difficile infections in the intensive care unit. The investigators hypothesize that this intervention will result in similar benefits outside of the intensive care unit, and so expanded the intervention to non-ICU medical and surgical wards. To increase the rigor of our program evaluation, the roll-out was conducted in a stepped-wedge randomized controlled design.

ELIGIBILITY:
All patients admitted to the medical/surgical services will be included in statistical analysis of program evaluation. The inclusion/exclusion criteria below, just define who receives the antibiotic stewardship intervention on each service.

Inclusion Criteria:

* admitted to one of these services: general internal medicine, cardiology, nephrology, orthopedic surgery, neurosurgery, general surgery or trauma surgery
* receiving 3rd or 10th day of treatment with one of the following antibiotics:
* ceftriaxone, ceftazidime, piperacillin-tazobactam, ciprofloxacin, levofloxacin, meropenem, ertapenem, vancomycin

Exclusion Criteria:

* patient being followed by the infectious diseases consult service

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19220 (Actual)
Dates: Start 2010-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Days of antibiotic therapy (DOTs) of targeted broadspectrum agents per patient days (PDs) | patients will be followed until discharge from hospital (expected median 7 days for those on antibiotics)
  * Targeted broadspectrum antibiotics include third generation cephalosporins (ceftriaxone, ceftazidime), beta-lactam beta-lactamase inhibitors (piperacillin-tazobactam), fluoroquinolones (ciprofloxacin, levofloxacin), carbapenems (ertapenem and meropenem), and glycopeptides (vancomycin)
  * DOTs are defined as the number of unique antibiotic agents prescribed each day (regardless of dose)

SECONDARY OUTCOMES:
Days of antibiotic therapy of any antibiotic agent(DOTs)per patient days (PDs) | patients will be followed until discharge from hospital (expected median 7 days for those on antibiotics)
  -Definition as per primary outcome, but can include any antibiotic (not just those broadspectrum agents targeted by the intervention)
Costs of antibiotic therapy ($) per patient day | patients will be followed until discharge from hospital (expected median 7 days for those on antibiotics)
  Based on acquisition costs for each agent.
Hospital-acquired Clostridium difficile infection. | patients will be followed until discharge from hospital (expected median 7 days for those on antibiotics)
  Cases of Clostridium difficile infection deemed to have been acquired during the current hospital stay by prospective Infection Prevention & Control surveillance team.
Antibiotic susceptibility of gram negative bacterial isolates | patients will be followed until discharge from hospital (expected median 7 days for those on antibiotics)

CONTACTS AND LOCATIONS:
Overall Officials: Nick Daneman, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] Elligsen M, Walker SA, Simor A, Daneman N. Prospective audit and feedback of antimicrobial stewardship in critical care: program implementation, experience, and challenges. Can J Hosp Pharm. 2012 Jan;65(1):31-6. doi: 10.4212/cjhp.v65i1.1101. No abstract available. PMID 22479110
- [Background] Elligsen M, Walker SA, Pinto R, Simor A, Mubareka S, Rachlis A, Allen V, Daneman N. Audit and feedback to reduce broad-spectrum antibiotic use among intensive care unit patients: a controlled interrupted time series analysis. Infect Control Hosp Epidemiol. 2012 Apr;33(4):354-61. doi: 10.1086/664757. PMID 22418630